CLINICAL TRIAL: NCT06919029
Title: Assessing the Effect of Advanced Hybrid Closed Loop System, MiniMed 780G With GS4 Glucose Sensor in Newly Diagnosed Children and Adolescents With Type 1 Diabetes on Glycemic Control and Patient Reported Outcomes Compared to Standard Insulin Therapy Historical Data (AHCL in New Onset T1D Children Study): a Single Arm Open- Label Prospective Observational Study Protocol
Brief Title: Effect of Advanced Hybrid Closed Loop System, MiniMed 780G in Newly Diagnosed Children and Adolescents With Type 1 Diabetes on Glycemic Control and Patient Reported Outcomes Compared to Standard Insulin Therapy Historical Data (AHCL in New Onset T1D Children Study)
Status: Recruiting | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Aghia Sophia Children's Hospital of Athens (Other)
Responsible Party: Principal Investigator, Christina Kanaka-Gantenbein, Professor Pediatrics- Pediatric Endocrinology, Director First Department of Pediatrics, National and Kapodistrian University of Athens, Medical School, "Aghia Sophia" Children's Hospital, National and Kapodistrian University of Athens
Other Study IDs: 6267/14.3.2025
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type I
Keywords: type 1 diabetes; advanced hybrid closed loop; diabetes onset
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Advanced Hybrid Closed Loop from onset of type 1 diabetes in children — The objective of this study is to evaluate glycemic control of users of the AHCL system MiniMed 780G with GS4 calibration-free sensor in children and adolescents with newly diagnosed T1D implemented directly upon T1D diagnosis in combination with continuous glucose monitoring system (CGMS) compared with those treated with MDI retrieved from historical data- in a single- arm open-label prospective observational study, assessed at 3 months. After the initial study period there will be a 3month extension phase of the study.

SUMMARY:
The objective of this study is to evaluate glycemic control of users of the AHCL system MiniMed 780G with GS4 calibration-free sensor in children and adolescents with newly diagnosed T1D implemented directly upon T1D diagnosis in combination with continuous glucose monitoring system (CGMS) compared with those treated with MDI retrieved from historical data- in a single- arm open-label prospective observational study, assessed at 3 months. After the initial study period there will be a 3month extension phase of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes (WHO criteria). Diagnosis of type 1 diabetes is based on international criteria and the investigator's judgment; C peptide level and antibody determinations are not required.
2. Age range 7 to 17 years.
3. Literate in Greek or English.
4. Willing to wear study devices.
5. Willing to follow study-specific instructions.
6. Total daily insulin dose greater than 8.0 units over 1 week period
7. Willing and able (access to internet from home) to download information into the Medtronic CareLink software
8. Clinically eligible to start the AHCL system

Exclusion Criteria:

* Type 2 diabetes mellitus or MODY diabetes
* Any untreated comorbidities of type 1 diabetes
* Medication affecting metabolic control or interfering in the interpretation of HbA1c
* Pregnancy
* Untreated diabetes retinopathy, or other causes that in the investigator's opinion, precludes the individual from participating in the trial.
* Known or suspected allergy to insulin.
* Regular use of acetaminophen.
* Lack of reliable telephone facility for contact.
* Living alone.
* Severe visual or hearing impairment.
* Medically documented allergy to the adhesive of plasters or unable to tolerate tape adhesive around sensor placement.
* Serious skin lesions at areas of the body used for insertion of the glucose sensor.
* Illicit drugs abuse.
* Alcohol abuse.
* Sickle cell disease, haemoglobinopathy, receiving red blood cell transfusion or erythropoietin within 3 months prior to time of enrollment.
* Eating disorder including anorexia/bulimia.
* Milk protein allergy.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study is a single-center open-label, single arm, trial, comparing advanced hybrid closed-loop (AHCL) insulin delivery and standard insulin therapy with multiple daily injections (MDI) (historical data- control) over a period of 3 months in newly diagnosed type 1 diabetes children and adolescents hospitalized and followed at the Diabetes center of the First Department of Pediatrics of the Medical School of the National and Kapodistrian University of Athens, Athens, Greece. After the initial 3 months, there will be an extension phase of the study, for another 3 months (total 6 months).
  A total of 30-35 individuals (aged 7-17 years) will be enrolled to reach 25-30 individuals who will complete the 3-months' study. The expected number of participants is based on the last 3 years data of our Diabetes Center, where the total number of newly diagnosed children/ adolescents with T1D (and those over 7 years of age) in our Center was as follows, in 2022: 56 (36), in 2023: 63 (47), in 2024.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
CGMS metrics | 3 and 6 months (extension phase)
  CGMS metrics including Time in Range (70-180 mg/dl) during the 3 months' study period, i.e. from baseline to 3 months (90 days) extracted from the CGMS data from both the study group and children and adolescents in MDI- FGM/CGM group (historical data from age and sex matched children and adolescents followed in the same Diabetes Center). The same metrics will be evaluated in the extension phase of the study, namely at 6-months post initiation of the study.
HbA1c | 3 months and 6 months (extension phase)
  HbA1c

SECONDARY OUTCOMES:
Acceptance of AHCL | 3 months
  Assess the percentage of the study participants willing to continue their therapy with AHCL as shown by prescribing the 780G insulin pump after the 3 months' time of their participation to the study.
TAR (Time Above Range) (>180mg/dl) | 3 months and 6 months (extension phase)
  Time Above Range (>180mg/dl) from baseline to 3 months (90 days) extracted from the CGMS data from both the study group and children and adolescents in MDI- FGM/CGM group (historical data from age and sex matched children and adolescents followed in the same Diabetes Center). The same metrics will be evaluated in the extension phase of the study, namely at 6-months post initiation of the study.
TBR (Time Below Range) (<70mg/dl) | 3 and 6 months (extension phase)
  TBR (Time Below Range) during the 3 months' study period, i.e. from baseline to 3 months (90 days) extracted from the CGMS data from both the study group and children and adolescents in MDI- FGM/CGM group (historical data from age and sex matched children and adolescents followed in the same Diabetes Center). The same metrics will be evaluated in the extension phase of the study, namely at 6-months post initiation of the study.
AHCL use | 3 and 6 months (extension phase)
  Advanced Hybrid Closed Loop use during the 3 months' study period, i.e. from baseline to 3 months (90 days) extracted from AHCL data. The same metric will be evaluated in the extension phase of the study, namely at 6-months post initiation of the study.
Total daily insulin requirements | 3 and 6 months (extension phase)
  Total daily insulin requirements during the 3 months' study period, i.e. from baseline to 3 months (90 days) extracted from the CGMS data from both the study group and children and adolescents in MDI- FGM/CGM group (historical data from age and sex matched children and adolescents followed in the same Diabetes Center). The same metrics will be evaluated in the extension phase of the study, namely at 6-months post initiation of the study.
Hypoglycemia Fear Survey for Children and Parents (HFS-C & P) | baseline, 3 months and 6 months (extension phase)
  QoL of the study participants before, 3 months and 6 months after initiation of the study, with the use of the questionnaire "Hypoglycemia Fear Survey for Children and Parents (HFS-C & P)"
PedsQL 3.0 Diabetes Module [Child (8-12 years of age) and Parent-Proxy Report for Children (ages 8-12), Adolescent (13-18 years of age), where appropriate | baseline, 3 months and 6 months (extension phase)
  QoL of the study participants before, 3 months and 6 months after initiation of the study, with the use of questionnaire "PedsQL 3.0 Diabetes Module [Child (8-12 years of age) and Parent-Proxy Report for Children (ages 8-12), Adolescent (13-18 years of age), where appropriate
Brief Illness Perception Questionnaire | baseline, 3 months and 6 months (extension phase)
  QoL of the study participants before, 3 months and 6 months after initiation of the study, with the use of questionnaire "Brief Illness Perception Questionnaire"
Fasting c-peptide, ΒΜΙ-SDS from baseline to 3 and 6 months | baseline, 3 months and 6 months (extension phase)
  Assess the change in fasting c-peptide from baseline to 3 and 6 months
ΒΜΙ-SDS | baseline, 3 months and 6 months (extension phase)
  Assess the change in ΒΜΙ-SDS from baseline to 3 and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- First Department of Pediatrics, National and Kapodistrian University of Athens, Medical School, "Aghia Sophia" Children's Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ware J, Boughton CK, Allen JM, Wilinska ME, Hartnell S, Thankamony A, Randell T, Ghatak A, Besser REJ, Elleri D, Trevelyan N, Campbell FM, Sibayan J, Bailey R, Calhoun P, Dunseath G, Hovorka R; CLOuD Consortium. Effect of 48 Months of Closed-Loop Insulin Delivery on Residual C-Peptide Secretion and Glycemic Control in Newly Diagnosed Youth With Type 1 Diabetes: A Randomized Trial. Diabetes Care. 2024 Aug 1;47(8):1441-1448. doi: 10.2337/dc24-0360. PMID 38924772
- [Background] Michaels VR, Boucsein A, Watson AS, Frewen CM, Sanders OJ, Haszard JJ, Jones SD, Milford-Hughes PJ, de Bock MI, Wheeler BJ. Glucose and Psychosocial Outcomes 12 Months Following Transition from Multiple Daily Injections to Advanced Hybrid Closed Loop in Youth with Type 1 Diabetes and Suboptimal Glycemia. Diabetes Technol Ther. 2024 Jan;26(1):40-48. doi: 10.1089/dia.2023.0334. Epub 2023 Nov 7. PMID 37823890
- [Background] Petrovski G, Al Khalaf F, Campbell J, Day E, Almajaly D, Hussain K, Pasha M, Umer F, Hamdan M, Khalifa A. Glycemic outcomes of Advanced Hybrid Closed Loop system in children and adolescents with Type 1 Diabetes, previously treated with Multiple Daily Injections (MiniMed 780G system in T1D individuals, previously treated with MDI). BMC Endocr Disord. 2022 Mar 29;22(1):80. doi: 10.1186/s12902-022-00996-7. PMID 35351095
- [Background] Boucsein A, Watson AS, Frewen CM, Sanders OJ, Haszard JJ, Jones SD, Milford-Hughes PJ, de Bock MI, Wheeler BJ. Impact of Advanced Hybrid Closed Loop on Youth With High-Risk Type 1 Diabetes Using Multiple Daily Injections. Diabetes Care. 2023 Mar 1;46(3):628-632. doi: 10.2337/dc22-1971. PMID 36689621